CLINICAL TRIAL: NCT06744270
Title: Inonu University Clinical Research Ethics Committee
Brief Title: Comparison of the Effects of Injectable Platelet-rich Fibrin and Low-dose Laser Applications on Palatal Wound Healing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esra Bozkurt (Other)
Collaborators: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Sponsor-Investigator, Esra Bozkurt, Assistant Professor Dr., Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024/83
Record Dates: First submitted 2024-12-15; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: Free gingival graft; Injectable platelet-rich fibrin; low-dose laser therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): The group in which no procedure was performed on the palatal wound area after free gingival grafting
- i-PRF group (Experimental): Immediately after the SDG operation, the venous blood taken from the patient will be centrifuged for 3 minutes at 2300 rpm in a centrifuge (PC-O2, Process for PRF, Nice, France) and two layers will be obtained: the lower layer is red blood cells and the upper layer is i-PRF. The i-PRF in the upper part of the tube will be collected with a syringe and transferred to the metal godet. 20-25 minutes will be waited for polymerization. After polymerization, the polymerized i-PRF will be applied to the wound surface in the donor area.
  Interventions: Other: i-PRF group
- low-dose laser group (Experimental): In the laser group, low-dose laser will be applied to the palatal donor area immediately after the FGG operation, on the 3rd, 5th, 7th and 14th days.
  Interventions: Other: low-dose laser group

INTERVENTIONS:
Other: i-PRF group — In the i-PRF group, 10 ml of venous blood taken from the patient immediately after the SDG operation will be transferred to a tube that does not contain any anticoagulant. The collected venous blood will be centrifuged for 3 minutes at 2300 rpm in a centrifuge device and two layers will be obtained: the lower layer is red blood cells and the upper layer is i-PRF. 20-25 minutes will be waited for polymerization. After polymerization, the polymerized i-PRF will be applied to the wound surface in the donor area. Following the operation, patients will be called for check-ups on the 3rd, 5th, 7th, 14th, 21st and 30th days and their photographs will be taken and the following parameters will be evaluated.
  * Pain assessment and analgesic intake
  * H2O2 Foaming Test (to assess epithelialization)
  * Wound healing will be assessed using the Image program from patient photographs
  * Edema and erythema scores will be assessed visually.
  Arms: i-PRF group
Other: low-dose laser group — In the laser group, low-dose laser will be applied to the palatal donor area immediately after SDG surgery, on the 3rd, 5th, 7th and 14th days. A GaAlAs diode laser (CHEESETM, GIGAA Laser, Wuhan Gigaa Optronics Technology Co., Ltd., China) with a wavelength of 810 nm and a low-dose diode laser application tip with a fiber diameter of 950 µm will be used. A low-dose diode laser will be applied to the surgical operation area in accordance with the manufacturer's instructions, with a non-contact regional 0.3 W power and an intensity of 4 J/cm2 in continuous mode for 1 min. Following the operation, patients will be called for check-ups on the 3rd, 5th, 7th, 14th, 21st and 30th days, and their photographs will be taken and the following parameters will be evaluated. • Pain assessment and analgesic intake
  * H2O2 Foaming Test (to assess epithelialization)
  * Wound healing will be assessed using Image program from patient photographs
  * Edema and erythema scores will be assessed visually.
  Arms: low-dose laser group

SUMMARY:
The investigators will evaluate the findings related to pain and bleeding, quality of life after surgery, and wound healing in participants who received injectable platelet-rich fibrin (i-PRF) and low-dose laser therapy to the palatal region after free gingival graft (FGG) surgery, compared to participants who did not receive any medication/active substance other than surgery. The investigators aim to evaluate whether i-PRF and low-dose laser treatments are superior to each other and to participants who did not receive any medication/active substance. The investigators predict that i-PRF and low-dose laser therapy will accelerate wound healing, reduce postoperative pain, and improve the patient's quality of life after surgery. The investigators do not expect any adverse effects from the application of i-PRF and low-dose laser therapy.

DETAILED DESCRIPTION:
Attached gingiva plays an important role in maintaining periodontal health. In the presence of insufficient attached gingiva, inflammation and root sensitivity, root caries and gingival recessions that cause esthetic complaints occur in periodontal tissues due to mucogingival stress in the relevant region and inadequate oral hygiene. In such cases, the width of insufficient attached gingiva should be increased with mucogingival periodontal plastic surgery procedures. Free gingival graft (FGG) is accepted as the most frequently used mucogingival surgical procedure to increase attached gingiva due to the predictability of the surgical result, simplicity of the technique and its applicability in wide operation areas including many teeth. In the FGG operation, a recipient bed is prepared in the region with insufficient attached gingiva. A free gingival graft containing epithelium and connective tissue is applied from the donor region in appropriate dimensions to this recipient bed. The palatal region is the most preferred donor area in terms of anatomical advantage, ideal tissue thickness and wide keratinized band harvest . The secondary wound formed in the donor area after FGG heals in 2-4 weeks and can cause many problems affecting patient comfort . Different products such as hemostatic agents, herbal products, ozonated oil, antibacterial and antiseptic agents, bioactive materials and platelet concentrates have been tested to accelerate wound healing and prevent these problems. Studies are ongoing to determine the product and method that provides optimal patient comfort and wound healing after surgery from these products known to have effects on wound healing.

Palatal donor area healing occurs with fibroblast proliferation, collagen synthesis, angiogenesis and wound contraction. Revascularization, immune system and epithelial cell proliferation are very important for optimal wound healing. It has been reported that platelet concentrates used in palatal wound healing accelerate wound healing and reduce postoperative patient discomfort by releasing growth factors such as transforming growth factor β (TGF-β), platelet-derived growth factor (PDGF), vascular endothelial growth factor (VEGF), and insulin-like growth factor-1 (IGF-1). Platelet-rich fibrin (PRF) has a three-dimensional fibrin network, and this structure and growth factor release enhance cell proliferation, migration, angiogenesis, and wound healing. The use of PRF in the palatal donor site after FGG surgery has been shown to provide significant benefits in terms of wound healing parameters and postoperative comfort. In recent years, there has been a need for an injectable formulation of PRF without the use of anticoagulants. This need was met with the introduction of a new platelet concentrate, Injectable platelet-rich fibrin (i-PRF), by Joseph Choukroun in 2014. I-PRF is obtained by centrifuging blood at low speed (700 rpm, 60 G). This concentrate is the injectable form of PRF and clots within a few minutes after injection. It is believed to contain not only white blood cells and platelets but also circulating stem cells and endothelial cells. Therefore, it is considered not only a platelet concentrate but also a "blood concentrate".

It has been reported that low-dose laser therapy has many areas of use in periodontal soft and hard tissues such as gingivitis, periodontitis, dentin sensitivity, gingivectomy and gingivoplasty, free gingival graft, guided tissue regeneration and peri-implantitis treatment and that it contributes positively to wound healing . The stimulating effects of low-dose laser therapy at the cellular level are based on the increase in blood flow in the damaged area and the formation of new capillaries, and faster healing of the tissue as a result of more oxygen supply. In addition, advantages such as increased cell respiration and Adenosine Triphosphate (ATP) synthesis, increased venous and lymphatic flow, collagen synthesis, anti-inflammatory effect and analgesic effect, stimulation of wound healing, immune system modulation, increased periodontal tissue attachment, increased bone regeneration, and reduced inflammatory status in periodontal pockets have been reported .

The investigators believe that the findings obtained as a result of the study will help determine the method that contributes the most to wound healing. Although there are many studies in the literature on low-dose laser and platelet concentrates in palatal wound healing, this study is the first to compare the contribution of 980 nm low-dose laser and i-PRF application to wound healing after FGG operations.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Systemically healthy,
* Not taking any medication that affects wound healing,
* Without clotting disorders or nausea,
* Patients who are not allergic to anti-inflammatory drugs.

Exclusion Criteria:

* Patients with systemic diseases (such as diabetes, hypertension, radiotherapy, chemotherapy),
* Patients who smoke or are active smokers and drink alcohol,
* Pregnant and breastfeeding women,
* Those with poor oral hygiene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 4 mounth
  The effects of i-PRF and low-dose laser groups on wound healing and patient quality of life will be evaluated statistically compared to each other and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Bozkurt, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sütçü İmam University, Faculty of Dentistry, Department of Periodontics, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We do not want to share study data

REFERENCES:
- [Background] Ozcan M, Ucak O, Alkaya B, Keceli S, Seydaoglu G, Haytac MC. Effects of Platelet-Rich Fibrin on Palatal Wound Healing After Free Gingival Graft Harvesting: A Comparative Randomized Controlled Clinical Trial. Int J Periodontics Restorative Dent. 2017 Sep/Oct;37(5):e270-e278. doi: 10.11607/prd.3226. PMID 28817141
- [Background] Kim SH, Tramontina VA, Papalexiou V, Luczsyzyn SM, De Lima AA, do Prado AM. Bismuth subgallate as a topical haemostatic agent at the palatal wounds: a histologic study in dogs. Int J Oral Maxillofac Surg. 2012 Feb;41(2):239-43. doi: 10.1016/j.ijom.2011.12.002. Epub 2011 Dec 29. PMID 22209184
- [Background] Ustaoglu G, Ercan E, Tunali M. The role of titanium-prepared platelet-rich fibrin in palatal mucosal wound healing and histoconduction. Acta Odontol Scand. 2016 Oct;74(7):558-564. doi: 10.1080/00016357.2016.1219045. Epub 2016 Aug 19. PMID 27538770
- [Background] Wang HL, Bunyaratavej P, Labadie M, Shyr Y, MacNeil RL. Comparison of 2 clinical techniques for treatment of gingival recession. J Periodontol. 2001 Oct;72(10):1301-11. doi: 10.1902/jop.2001.72.10.1301. PMID 11699470
- [Background] Wennstrom J, Pini-Prato G. Mucogingival therapy-periodontal plastic surgery. In: Lindhe J, Karring T, Lang N (eds). Clinical Periodontlogy and Implant Dentistry, 4th ed. Oxford, Blackwell Munksgaard, 2003: 588-92
- [Background] Newman MG, Takei H, Klokkevold PR, Carranza FA. Carranza's Clinical Periodontology, 12th ed. St. Louis, Missouri, 2012.
- [Derived] Bozkurt E, Ozdemir EC. The efficacy of injectable platelet-rich fibrin versus photobiomodulation therapy on palatal wound healing: a randomized, controlled, clinical trial. Clin Oral Investig. 2025 Oct 15;29(11):512. doi: 10.1007/s00784-025-06613-w. PMID 41091419
- See also: Inonu University Clinical Research Ethics Committee — https://www.inonu.edu.tr/klinik.etik
- Available data/document: Clinical Study Report: Inonu University Clinical Rese — https://www.inonu.edu.tr/klinik.etik — https://www.inonu.edu.tr/klinik.etik